CLINICAL TRIAL: NCT01862601
Title: Study to Evaluate the Safety and Performance of the JetTouch Needle-Free Endoscopic Injection System to Deliver Saline Into the Bladder Wall of Healthy Subjects
Brief Title: JetTouch Injection System to Deliver Saline Into the Bladder Wall of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Medical Systems (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OT1202
Record Dates: First submitted 2013-05-20; First posted 2013-05-24 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JetTouch injections (Experimental)
  Interventions: Device: JetTouch Needle-free injection system

INTERVENTIONS:
Device: JetTouch Needle-free injection system — Needle-free injection system believed to provide consistent and reliable delivery of material to the bladder wall.

SUMMARY:
This research study is being done to see how well the JetTouch Needle-Free Endoscopic Injection System is able to deliver a solution safely into the bladder wall. The JetTouch Needle-Free Endoscopic Injection System is a jet injector that allows fluids to be injected into the bladder without using a needle. It is hoped that this method will provide a reliable and consistent method to deliver drugs into the bladder wall.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (male and female) aged 18-55 without urinary complaints or documented urinary tract dysfunctions.

Exclusion Criteria:

* Unable or unwilling to sign Informed Consent Form or comply with study requirements
* Non-English speaking
* Currently enrolled in another clinical trial
* Undergone treatments given into the bladder in the past 4 weeks
* Female subject and has a positive urine pregnancy test at the time of screening/procedure or intends to become pregnant while enrolled
* Female subject and is currently breast feeding
* Female subject and has given birth in past 6 months
* Current or history of chronic urinary tract infections
* Current or history of chronic hematuria
* Current or history of bladder cancer
* History of major surgery in the last 6 months
* Current or history of bleeding disorders
* Currently taking anticoagulants
* Taking aspirin and is unable to discontinue treatment for 2 weeks prior to bladder injection
* Taking NSAIDS and is unable to discontinue 48 hours prior to bladder injection
* Platelet count, prothrombin time/INR (PT/INR) and partial thromboplastin time (PTT) outside the normal limits of the laboratories established reference ranges
* Current or history of any of the following: neurogenic bladder, radiation to pelvic area, inflammation of the bladder wall because of tuberculosis, schistosomiasis, bladder or ureteric calculi
* Known hypersensitivity to any of the agents used in the injection (FLEXLINE-Bladder® Attachment material, lidocaine, saline, Indigo Carmine dye or Ciprofloxacin)
* Current or history of any medical condition that in the opinion of the Investigator would make them an unsuitable candidate for this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety of the JetTouch system to deliver saline into the bladder wall. | within 14 days of the JetTouch procedure
Ability of the JetTouch system to deliver saline into the bladder wall. | At the JetTouch procedure

SECONDARY OUTCOMES:
Physician feedback on the use of the JetTouch system. | At the JetTouch Procedure
Physician feedback on perceived subject tolerability of the JetTouch injection procedure. | At the JetTouch procedure.
Subject feedback question regarding the procedure. | At the JetTouch procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Chapple, BSc MD DHC FRCS (Urol) FEBU, Principal Investigator — Consultant Urological Surgeon, Royal Hallamshire Hospital
Locations (2):
- United Kingdom (2):
  - Guy's Hospital / Quintiles, Ltd., London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield